CLINICAL TRIAL: NCT03125239
Title: A Phase 1 Study of Merestinib in Combination With LY2874455 in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Combination Merestinib and LY2874455 for Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jacqueline Garcia, MD (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Jacqueline Garcia, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-099
Record Dates: First submitted 2017-04-17; First posted 2017-04-24 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Relapsed Adult Acute Myeloid Leukemia; Refractory Adult Acute Myeloid Leukemia
Keywords: Refractory Adult Acute Myeloid Leukemia; Relapsed Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — merestinib; 2-(4-(2-(5-(1-(3,5-dichloropyridin-4-yl)ethoxy)-1H-indazol-3yl)vinyl)-1H-pyrazol-1-yl)ethanol

STUDY DESIGN:
Intervention Model Description: open-label phase 1 study using a 3+3 design with planned dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Merestinib and LY2874455 (Experimental): Patients who fulfill eligibility criteria will be entered into the trial to receive Merestinib and LY2874455.
  After the screening procedures confirm participation in the research study:
  * The investigators are looking for the highest dose of the combination of study drugs that can be administered safely without severe or unmanageable side effects in participants that have AML, not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.
  * Merestinib
  * LY2874455
  Interventions: Drug: Merestinib; Drug: LY2874455

INTERVENTIONS:
Drug: Merestinib — Oral, once a day, Merestinib Only- Lead in period on week. The followed by cycles on combination therapy with Merestinib and LY2874455 (28 days long)
  Other Names: LY2801653
Drug: LY2874455 — This will be followed by cycles of combination therapy with merestinib and LY2874455. Each of these cycles are 28 days long. • LY2874455 will be taken by mouth twice a day. You may take LY2874455 twice daily for 14 days, 21 days, or 28 days each cycle depending on the dose level you are assigned.

SUMMARY:
This research study is studying a combination of two targeted therapies as a possible treatment for acute myeloid leukemia (AML) that has relapsed after initial treatment or did not fully respond.

The name of the study interventions involved in this study are:

* Merestinib
* LY2874455

DETAILED DESCRIPTION:
* This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.
* The FDA (the U.S. Food and Drug Administration) has not approved Merestinib or LY2874455 as a treatment for any disease.
* Merestinib is an oral drug known as a MET kinase inhibitor that is being developed as a treatment for patients with advanced cancer. MET inhibitors work by stopping a signal that a cell receives instructing it to grow.
* LY2874455 is an oral drug known as an FGFR inhibitor that is also being developed as a treatment for patients with advanced cancer. FGFR inhibitors work by stopping a signal that a cell receives instructing it to grow.
* In this research study, the investigators are investigating whether Merestinib and LY2874455 is safe to give in combination in patients with AML. In previous laboratory studies, it was found that leukemia cells responded to treatment with a MET inhibitor and an FGFR inhibitor. However, it is not yet known whether this will also be the case with LY2874455 and merestinib when given to participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed relapsed or refractory acute myeloid leukemia (AML) or secondary AML following IWG criteria [40].

  * For subjects with relapsed AML: evidence of ≥ 5% blasts in the bone marrow or development of extramedullary disease who relapse after:

    * Allogeneic hematopoietic stem cell transplant, or
    * A minimum of one cycle of standard cytotoxic chemotherapy or two cycles of any hypomethylating agent-based therapy
  * For subjects with refractory AML: a minimum of 2 prior induction regimens (example: patients who receive 7+3 followed by 5+2 would count as one induction regimen) or a minimum of two cycles of any hypomethylating agent-based therapy.
  * For subjects with secondary AML: untreated secondary AML, must have been previously treated for myelodysplastic syndrome (MDS) or myeloproliferative neoplasms (MPN) or MDS/MPN (MDS/MPN) overlap syndrome.
* No limit to number of prior therapies.
* Patients are considered to have failed available therapies or to be ineligible for or to not be interested in intensive chemotherapies, including allogeneic hematopoietic stem cell transplantation.
* Patients with a history of allogeneic stem cell transplantation are eligible for study participation provided the transplant was > 100 days prior to study enrollment. Patients must not have active graft versus host disease other than grade 1 skin involvement.
* Age 18 and older.
* ECOG performance status ≤2 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * Direct bilirubin within ≤ 1.5 times the institutional upper limit of normal (ULN). For patients with known Gilbert Syndrome, or if the elevation is believed to be leukemia related, the cut-off of ≤ 3.0 times the institutional ULN is allowable.
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN, unless believed to be leukemia related then ≤ 5 x ULN is allowed.
  * Serum creatinine ≤ 2.0 x ULN
* Females of child bearing potential and males must agree to use barrier method/hormonal methods from start of study until four months after last dose of study drug. Females of child bearing potential must have a negative serum pregnancy test at screening. Females are not considered to be of child bearing potential if they are status post successful surgical sterilization including hysterectomy, bilateral tubal ligation or bilateral oophorectomy, or if they are postmenopausal (absence of menses for 12 consecutive months that is not secondary to prior chemotherapy, anti-estrogens, ovarian suppression or other reversible cause).
* The effects of Merestinib and LY2874455 on the developing human fetus are unknown. Small molecular inhibitors of tyrosine kinase receptors are known to be teratogenic. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Able and willing to undergo the required bone marrow biopsies. Correlative studies are strongly encouraged.

Exclusion Criteria:

* Participants who have had radiotherapy within 2 weeks, with the exception of localized radiotherapy to palliate extramedullary leukemia where no washout is required.
* Participants who have had chemotherapy within 2 weeks or 5 half-lives (whichever is longer) from the last dose of chemotherapy prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Hydroxyurea is allowed per treating investigator. IT chemotherapy prophylaxis is permitted.
* Participants who are receiving any other investigational agents, with the exception of topical or ophthalmologic therapies for mild graft versus host disease which are permitted.
* Participants with known CNS leukemia involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Individuals with other active malignancies that require concurrent chemotherapy are ineligible. Hormone therapy is allowed.
* Subject has a known gastrointestinal disorder that in the opinion of the treating investigator is concerning for malabsorption of oral medications.
* Subject is unable to swallow pills.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients with current or history of NYHA class III or IV cardiac disease, myocardial infarction with past 6 months, or unstable arrhythmia will be ineligible for study.
* Pregnant women are excluded from this study because Merestinib and LY2874455 have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Merestinib and LY2874455, breastfeeding should be discontinued if the mother is treated with Merestinib and LY2874455.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Merestinib and LY2874455. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Subjects with QTcF interval of ≥ 450 msec if male and ≥ 470 msec if female following or with other factors increase the risk of QT prolongation or arrhythmic events (e.g. heart failure, hypokalemia, family history of long QT interval syndrome) at screening. Subjects with bundle branch block should be reviewed by the Medical Monitor for potential inclusion.
* Subjects with known active HBV or HCV (cannot have an elevated viral load of HBV or HCV if known history) are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
MTD of LY2874455 and Merestinib | 35 Days
  Dose-escalation will follow a standard 3+3 design exploring 3 dose levels of LY2874455 with a steady dose of Merestinib. We will escalate to next dose cohort if 0/3 or 1/6 participants have a DLT during the first cycle of therapy. If the rate of dose limiting toxicity (DLT) exceeds 30%, it is less likely that the dose of LY2874455 will be escalated.

SECONDARY OUTCOMES:
Best Overall response | Up to 1 year
  Time to event summaries will use the Kaplan-Meier method.
Duration of Remission | Up to 1 year
  Time to event summaries will use the Kaplan-Meier method.
Progression Free Survival | Up to 1 year
  Time to event summaries will use the Kaplan-Meier method.
Overall Survival | Up to 1 year
  Time to event summaries will use the Kaplan-Meier method.
PK of Merestinib and LY2874455 in AML during the dose escalation part of the study: AUC | 35 days
  Standard noncompartmental pharmacokinetic analysis will be employed including AUC 0-24 after initial and repeat administration.
PK of Merestinib and LY2874455 in AML during the dose escalation part of the study: Cmax | 35 days
  Standard noncompartmental pharmacokinetic analysis will be employed including peak drug plasma concentration (Cmax) after initial and repeat administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline S. Garcia, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts